CLINICAL TRIAL: NCT03268330
Title: Role of Macrophage Migratory Inhibitory Factor in Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naima eid, Principal investigator, Assiut University
Other Study IDs: ROMMIFISS
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: System; Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Migration Inhibitory Factor has proliferative and antiapoptotic actions on fibroblasts which may be relevant to scleroderma because of the central role of a dysregulated fibroproliferative response in disease-affected tissues

DETAILED DESCRIPTION:
* Systemic sclerosis (scleroderma) is a disease of unknown etiology characterized by fibrosis of the skin and internal organs, pronounced vasculopathy, and dysregulated immune system.
* Clinically, the disease is divided into 2 major subsets, diffuse cutaneous SSc (dcSSc) and limited cutaneous SSc (lcSSc). The diffuse cutaneous subtype is generally associated with significant internal organ involvement, especially renal crisis and diffuse alveolitis of the lung, along with antitopoisomerase (antitopo) autoantibody. The limited cutaneous subtype is distinguished by Raynaud's phenomenon, telangiectasias, pulmonary hypertension, and the presence of anticentromere antibody. However, there is significant overlap both in the clinical manifestations and in the specific autoantibodies that occur in these subtypes. It is not known what predisposes a susceptible individual to develop one subtype versus another, nor is there significant information about how the 2 disease subtypes may be pathogenically related.
* Activation of T lymphocytes and macrophages is an early event in the parthenogenesis of SSc. Activated T cells , macrophages and endothelial cells are important sources of Macrophage Migration Inhibitory Factor MIF was initially identified as the protein secreted by activated T lymphocytes capable of inhibiting random migration of macrophages, concentrating macrophages at inflammation loci, and enhancing their ability to kill intracellular parasites and tumoral cells.
* Migration Inhibitory Factor has proliferative and antiapoptotic actions on fibroblasts which may be relevant to scleroderma because of the central role of a dysregulated fibroproliferative response in disease-affected tissues.
* In patients with SSc, elevated serum levels of MIF, increased MIF expression in the skin and afunctional promoter polymorphism in the MIF gene that might influence clinical expression have been described therefore MIF might have an important role in the disease.

ELIGIBILITY:
Inclusion Criteria:

-Patients with Systemic Sclerosis .

Exclusion Criteria:

* Patients with Interstitial Pulmonary Fibrosis caused by causes other than SSc.
* Other rheumatologic diseases.
* Overlap or Mixed diseases.
* Patients with renal disease caused by causes other than SSc.
* Unwillingness to participate in the study.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -Patients with Systemic Sclerosis diagnosed by Rheumatologists at Department of Rheumatology, Rehabilitation and Physical Medicine Assiut University.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between Migration Inhibitory Factor and some of the clinical manifestations of Systemic Sclerosis. | 1 hour
  Serum levels of Macrophage Migratory Inhibitory Factor will be measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Doaa K Mohamed, Lectruer, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assiut University Hospital, Asyut
  - Assuit University hospital, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sakkas LI, Chikanza IC, Platsoucas CD. Mechanisms of Disease: the role of immune cells in the pathogenesis of systemic sclerosis. Nat Clin Pract Rheumatol. 2006 Dec;2(12):679-85. doi: 10.1038/ncprheum0346. PMID 17133253
- [Background] Selvi E, Tripodi SA, Catenaccio M, Lorenzini S, Chindamo D, Manganelli S, Romagnoli R, Ietta F, Paulesu L, Miracco C, Cintorino M, Marcolongo R. Expression of macrophage migration inhibitory factor in diffuse systemic sclerosis. Ann Rheum Dis. 2003 May;62(5):460-4. doi: 10.1136/ard.62.5.460. PMID 12695161
- [Background] Wu SP, Leng L, Feng Z, Liu N, Zhao H, McDonald C, Lee A, Arnett FC, Gregersen PK, Mayes MD, Bucala R. Macrophage migration inhibitory factor promoter polymorphisms and the clinical expression of scleroderma. Arthritis Rheum. 2006 Nov;54(11):3661-9. doi: 10.1002/art.22179. PMID 17075815
- [Background] Mitchell RA, Metz CN, Peng T, Bucala R. Sustained mitogen-activated protein kinase (MAPK) and cytoplasmic phospholipase A2 activation by macrophage migration inhibitory factor (MIF). Regulatory role in cell proliferation and glucocorticoid action. J Biol Chem. 1999 Jun 18;274(25):18100-6. doi: 10.1074/jbc.274.25.18100. PMID 10364264
- [Background] Calandra T, Bernhagen J, Mitchell RA, Bucala R. The macrophage is an important and previously unrecognized source of macrophage migration inhibitory factor. J Exp Med. 1994 Jun 1;179(6):1895-902. doi: 10.1084/jem.179.6.1895. PMID 8195715